CLINICAL TRIAL: NCT07355699
Title: Application of Orelabrutinib With or Without CD20 Monoclonal Antibody in Previously Untreated Marginal Zone Lymphoma:A Phase II, Prospective, Multicenter, Single-Arm Clinical Study
Brief Title: Application of Orelabrutinib With or Without CD20 Monoclonal Antibody in Previously Untreated Marginal Zone Lymphoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, LIANG WANG, Chief Physician of Hematology Department, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TREC2025-KY209
Record Dates: First submitted 2025-11-20; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Marginal Zone Lymphoma(MZL)
Keywords: Marginal Zone Lymphoma; Orelabrutinib; CD20 Monoclonal Antibody
MeSH Terms: conditions — Lymphoma, B-Cell, Marginal Zone | interventions — orelabrutinib; Rituximab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib-based treatments (Experimental): This is a single-arm study without a control group. All subjects will receive orelabrutinib treatment but will be stratified based on disease stage and clinical characteristics into the following two groups:
  1. Stage I MZL Patient Group (Monotherapy Group) Treatment regimen: Orelabrutinib monotherapy. Dosage and administration: Orelabrutinib 150mg, once daily (qd), taken continuously for 21 days per treatment cycle (d1-d21), for a total of 6 cycles (C1-C6).
  2. Stage II-IV MZL Patient Group (Combination Therapy Group) Treatment regimen: Orelabrutinib combined with a CD20 monoclonal antibody. Dosage and administration: Orelabrutinib 150mg, once daily (qd), taken continuously for 21 days per treatment cycle (d1-d21), for a total of 6 cycles (C1-C6). CD20 monoclonal antibody (either Rituximab 375mg/m², intravenous infusion, Day 1 of each cycle, C1-C6; or Obinutuzumab 1000mg, intravenous infusion, on Days 1, 8, and 15 of Cycle 1 [C1], and on Day 1 of Cycles 2-6 [C2-C6].
  Interventions: Drug: Orelabrutinib

INTERVENTIONS:
Drug: Orelabrutinib — 1. Stage I MZL Patients:
     Treatment with Orelabrutinib monotherapy. Induction Phase: During Cycles 1-6 (C1-C6), Orelabrutinib 150mg is administered orally once daily (qd) on Days 1-21 (d1-d21) of each cycle.
  2. Stage II-IV MZL Patients:
  Treatment with the Orelabrutinib plus CD20 monoclonal antibody regimen, divided into an induction phase and a maintenance phase.
  Induction Phase: During Cycles 1-6 (C1-C6), Orelabrutinib 150mg is administered orally once daily (150mg qd d1-d21/C1-C6). Concurrently, a CD20 monoclonal antibody is used: either Rituximab 375mg/m² intravenously (iv) on Day 1 of each cycle (d1/C1-C6); or Obinutuzumab, administered as 1000mg intravenously on Days 1, 8, and 15 of Cycle 1 (1000mg iv d1,d8,d15/C1), followed by 1000mg intravenously on Day 1 of Cycles 2-6 (1000mg iv d1/C2-C6).
  Maintenance Phase: If maintenance therapy is administered, during Cycles 7-30 (C7-C30), Orelabrutinib 150mg is administered orally once daily (qd) on Days 1-28 (d1-d28) of each cycle.
  Other Names: Rituximab; Obinutuzumab

SUMMARY:
This study focuses on treatment-naïve marginal zone lymphoma (MZL) patients and aims to investigate the efficacy and safety of orelabrutinib combined with or without CD20 monoclonal antibody.

This is a single-arm study without a control group. All subjects will receive orelabrutinib treatment but will be stratified based on disease stage and clinical characteristics into the following two groups:

1. Stage I MZL Patient Group (Monotherapy Group) Treatment regimen: Orelabrutinib monotherapy. Dosage and administration: Orelabrutinib 150mg, once daily (qd), taken continuously for 21 days per treatment cycle (d1-d21), for a total of 6 cycles (C1-C6).

   Target population: Patients with Ann Arbor Stage I gastric MALT MZL, including H. pylori-negative patients or those with unsatisfactory response after anti-H. pylori therapy, as well as other Stage I MZL patients unsuitable for local radiotherapy.

   Sample size: 50 cases.
2. Stage II-IV MZL Patient Group (Combination Therapy Group) Treatment regimen: Orelabrutinib combined with a CD20 monoclonal antibody. Dosage and administration: Orelabrutinib 150mg, once daily (qd), taken continuously for 21 days per treatment cycle (d1-d21), for a total of 6 cycles (C1-C6). CD20 monoclonal antibody (either Rituximab 375mg/m², intravenous infusion, Day 1 of each cycle, C1-C6; or Obinutuzumab 1000mg, intravenous infusion, on Days 1, 8, and 15 of Cycle 1 [C1], and on Day 1 of Cycles 2-6 [C2-C6]).

Target population: Patients with Ann Arbor Stage II-IV non-gastric MALT MZL, nodal MZL, splenic marginal zone lymphoma (SMZL), and other Stage II-IV MZL patients unsuitable for local radiotherapy.

Sample size: 38 cases.

DETAILED DESCRIPTION:
This study focuses on treatment-naïve marginal zone lymphoma (MZL) patients and aims to investigate the efficacy and safety of orelabrutinib combined with or without CD20 monoclonal antibody. Given the current lack of a standard first-line treatment regimen for MZL, and the limited efficacy and significant side effects associated with commonly used immunochemotherapy regimens, chemotherapy-free approaches have attracted considerable attention. As a domestically developed new-generation BTK inhibitor, orelabrutinib exhibits high selectivity and a favorable safety profile, and demonstrates synergistic effects with CD20 monoclonal antibodies. The study enrolls treatment-naïve MZL patients at different stages, administering either orelabrutinib monotherapy or combination therapy with a CD20 monoclonal antibody. Efficacy indicators, such as overall response rate and complete response rate, are closely monitored, with tumor changes assessed through regular imaging and laboratory examinations. Meanwhile, all types of adverse reactions are documented in detail to evaluate safety. Long-term follow-up is conducted to track progression-free survival and overall survival, comprehensively analyzing whether this combination regimen can emerge as a highly effective, low-toxicity, chemotherapy-free option.

This is a single-arm study without a control group. All subjects will receive orelabrutinib treatment but will be stratified based on disease stage and clinical characteristics into the following two groups:

1. Stage I MZL Patient Group (Monotherapy Group) Treatment regimen: Orelabrutinib monotherapy. Dosage and administration: Orelabrutinib 150mg, once daily (qd), taken continuously for 21 days per treatment cycle (d1-d21), for a total of 6 cycles (C1-C6).

   Target population: Patients with Ann Arbor Stage I gastric MALT MZL, including H. pylori-negative patients or those with unsatisfactory response after anti-H. pylori therapy, as well as other Stage I MZL patients unsuitable for local radiotherapy.

   Sample size: 50 cases.
2. Stage II-IV MZL Patient Group (Combination Therapy Group) Treatment regimen: Orelabrutinib combined with a CD20 monoclonal antibody. Dosage and administration: Orelabrutinib 150mg, once daily (qd), taken continuously for 21 days per treatment cycle (d1-d21), for a total of 6 cycles (C1-C6). CD20 monoclonal antibody (either Rituximab 375mg/m², intravenous infusion, Day 1 of each cycle, C1-C6; or Obinutuzumab 1000mg, intravenous infusion, on Days 1, 8, and 15 of Cycle 1 [C1], and on Day 1 of Cycles 2-6 [C2-C6]).

Target population: Patients with Ann Arbor Stage II-IV non-gastric MALT MZL, nodal MZL, splenic marginal zone lymphoma (SMZL), and other Stage II-IV MZL patients unsuitable for local radiotherapy.

Sample size: 38 cases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Pathologically confirmed marginal zone lymphoma;
* Presence of evaluable lesions;
* Meets indications for treatment: Fulfills the GELF criteria OR has disease-related clinical symptoms/organ function impairment;
* Patients who are unsuitable for local radiotherapy, refuse local radiotherapy, or have disease progression after local therapy. Cases considered unsuitable for local radiotherapy include the following:

Gastric MALT MZL, Ann Arbor stage I, that is H. pylori-negative, or H. pylori-positive gastric MALT MZL (Ann Arbor stage I) with poor response to H. pylori eradication therapy;

Non-gastric MALT and nodal MZL in Ann Arbor non-contiguous stage II or stages III-IV;

SMZL;

Gastric MALT classified as Lugano II2, IIE, or IV stage;

Patient intolerance to radiotherapy;

Other MZL patients deemed unsuitable for local radiotherapy by the investigator.

* ECOG score of 0-3;
* Expected survival time ≥ 3 months;
* Ability to provide signed informed consent.

Exclusion Criteria:

* Currently diagnosed with another malignant tumor;
* Central nervous system involvement by lymphoma or transformation to a higher grade;
* Allergy to any of the investigational drugs;
* Active infection or uncontrolled HBV infection, HIV/AIDS, or other serious infectious diseases;
* Pregnancy, lactating women, or subjects of childbearing potential unwilling to use contraception;
* Other situations deemed by the investigator as unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | From enrollment to the end of treatment at 21 weeks
  Best Overall Response Rate (ORR): Efficacy is assessed every two treatment cycles. The best ORR achieved within the 6 treatment cycles serves as the primary endpoint.

SECONDARY OUTCOMES:
Complete Response Rate | From enrollment to the end of treatment at 21 weeks
  Best Complete Response Rate (CRR): Efficacy is assessed every two treatment cycles. The best CRR achieved within the 6 treatment cycles serves as a secondary endpoint.
2-Year Progression-Free Survival Rate | From enrollment to 2 years
  2-Year PFS (Progression-Free Survival) refers to the time interval from the date a patient begins treatment until either disease progression, relapse, or death from any cause reaches two years. If the patient does not experience disease progression and remains alive within the two-year period, they are considered to have achieved 2-year PFS. If disease progression or death occurs within the two years, 2-year PFS is not achieved.
2-Year Overall Survival Rate | From enrollment to 2 years
  2-Year Overall Survival Rate (OS): OS is defined as the time from the date of study enrollment until the patient dies from any cause or is lost to follow-up.
AE | Through study completion, an average of 2.5 years
  Safety is evaluated according to the CTCAE v5.0 criteria. Toxicity assessments are performed during each treatment cycle, primarily focusing on hematological toxicities and non-hematological toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Wang, MD, Principal Investigator — Beijing Tongren Hospital
Locations (3):
- China (3):
  - Beijing Tongren Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital of China Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Time Frame: after the publishment of this study
Access Criteria: upon request to the PI after the publishment of this study